CLINICAL TRIAL: NCT02718937
Title: A Randomised, Phase 2a, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Antiviral Activity Against Respiratory Syncytial Virus Infection, and the Pharmacokinetics of Multiple Oral Doses of BTA-C585 in the Virus Challenge Model
Brief Title: Safety, Efficacy and Pharmacokinetics of BTA-C585 in a RSV Viral Challenge Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biota Pharma Europe Limited (Industry)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTA585-003
Record Dates: First submitted 2016-03-21; First posted 2016-03-24 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Syncytial Virus (RSV) Infection
Keywords: Viral diseases; Antiviral; Paramyxoviridae infections; RSV; Aviragen Therapeutics, Inc.; Aviragen Therapeutics; Aviragen
MeSH Terms: conditions — Infections; Virus Diseases; Paramyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BTA-C585 (Experimental): BTA-C585 100 mg oral capsule
  Interventions: Drug: BTA-C585 oral capsule
- Placebo (Placebo Comparator): Matching placebo capsule
  Interventions: Drug: Matching placebo capsules

INTERVENTIONS:
Drug: BTA-C585 oral capsule
  Other Names: BTA585
  Arms: BTA-C585
Drug: Matching placebo capsules
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the antiviral activity of oral BTA-C585 compared to placebo in healthy volunteers after intranasal challenge with RSV-A Memphis 37b virus.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female
2. Between 18 to 50 years old
3. Body mass index of 18 to 30 kg/m2

Exclusion Criteria:

1. Acute or chronic medical illness
2. Abnormal lung function Positive for HIV, Hepatitis B or C
3. Any significant abnormality of the nose or nasopharynx

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) viral load of RSV-A Memphis 37b | Days 2-13

SECONDARY OUTCOMES:
Area under the curve (AUC) of total RSV symptom scores | Days 1-13
Number of adverse events | Screening to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Anna Novotney-Barry, Study Director — Aviragen Therapeutics, Inc.
Locations (1):
- Biota Investigational Site, London, United Kingdom